CLINICAL TRIAL: NCT02963883
Title: Erythrocyte Transfusion Based on the Measurement of Central Venous Oxygen Saturation in Postoperative Cardiac Surgery: a Bicentric, Prospective Randomized Study
Brief Title: Erythrocyte Transfusion Based on the Measurement of Central Venous Oxygen Saturation in Postoperative Cardiac Surgery
Acronym: PITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2016_843_0015
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery
Keywords: ScVO2; Post operative red cell transfusion
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SVO2 group (Experimental): After optimization of oxygenation and blood volume, concentrate transfusion (s) of red blood cells by the individual value of ScvO2, whose value must be greater than 70% after elimination of hypovolemia, hypotension or hypoxemia.
  Interventions: Other: SVO2 group / control group
- control group (Active Comparator): After optimization of oxygenation and blood volume, concentrate transfusion (s) of red blood cells based on the hemoglobin values, as recommended by the National Health Authority for Anesthesiology, Surgery, Emergency (November 2014 ): transfusion threshold of <9 g / dl for patients with cardiovascular antecedents.
  Interventions: Other: SVO2 group / control group

INTERVENTIONS:
Other: SVO2 group / control group

SUMMARY:
Postoperative erythrocytes transfusion is associated with morbidity and excess mortality, which should lead to ask the indication for RBC transfusions only on metabolic needs. Currently, the majority of studies used to put hemoglobin values indicating red cell transfusions. Two observational studies have confirmed that a transfusion strategy based on a metabolic index (ScvO2) individual was accompanied by a different transfusion strategy than using the hemoglobin threshold values. We propose to conduct the first randomized multicenter study to evaluate erythrocyte transfusion strategy in postoperative cardiac surgery using the ScvO2 each patient versus a threshold value usually recommended for all patients.

DETAILED DESCRIPTION:
Postoperative erythrocytes transfusion is associated with morbidity and excess mortality, which should lead to ask the indication for RBC transfusions only on metabolic needs. Currently, the majority of studies used to put hemoglobin values indicating red cell transfusions. Two observational studies have confirmed that a transfusion strategy based on a metabolic index (ScvO2) individual was accompanied by a different transfusion strategy than using the hemoglobin threshold values. We propose to conduct the first randomized multicenter study to evaluate erythrocyte transfusion strategy in postoperative cardiac surgery using the ScvO2 each patient versus a threshold value usually recommended for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years
2. programmed cardiac surgery
3. Central venous catheter placed in territory SVC
4. Affiliation to a social security system
5. Hemoglobin <9 g / dL (transfusion threshold retained by the recommendations the HAS in November 2014 for perioperative patients with cardiovascular antecedents)

Exclusion Criteria:

1. Patient minor or under court protection
2. Pregnant or lactating women
3. severe acute hemorrhagic syndrome (defined by bleeding rate greater than 1.5 ml / kg / hour for 6 consecutive hours and / or surgical revision within the first 24 postoperative hours)
4. Installation of an external or internal circulatory support
5. emergency surgery (<24 hours from admission)
6. Complex Aortic Surgery
7. Sepsis
8. Patient Refusal of transfusion (religious belief)
9. Patient under guardianship
10. Renal failure with dialysis treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Number of patients transfused | 15 dys
  Number of patients transfused at least one red blood cell concentrate in postoperative cardiac surgery for the ScvO2 group compared to the control group

SECONDARY OUTCOMES:
acute pulmonary edema due to the overload | 15 days
  acute pulmonary edema due to overload or TACO, defined as acute pulmonary edema overload confirmed by clinical examination and echocardiography and leading to medical treatment
lesional pulmonary edema or TRALI, | 6 h
  lesional pulmonary edema or TRALIassociating acute respiratory distress within 6 hours of transfusion, bilateral infiltrates on chest radiograph, but without respiratory or elevated left ventricular load conditions precedent to echocardiography, and possibly confirmed by tests biological HLA
myocardial infarction | 15 days
  myocardial infarction, defined by elevated serum troponin dosing greater than 10 times the 99th percentile associated with electrocardioscopic changes (appearance of new Q waves or left bundle branch block), ultrasound (appearance of segmental disorder myocardial kinetics) or angiographic (occlusion of a coronary artery or bypass surgery), as defined by the European society of cardiology in 2012,
stroke | 15 days
  stroke, defined by a computed tomography documentation
acute renal failure, | 15 days
  acute renal failure, defined as an increase of at least 50% and / or 26.5 micromol / l of postoperative serum creatinine with respect to the preoperative baseline value and / or urine output less than 0.5 mL / kg / hr about 6 hours (definition of the international society of nephrology KDIGO)
immunological complications including allo-immunization | 15 days
  immunological complications including allo-immunization, immunological incompatibility and hemolytic accidents involving clinical symptoms (chills, fever, back pain), increased serum bilirubin, decreased the haptoglobinemy the positivization direct antiglobulin test ( DAT), or even looking for irregular antibodies as well as disseminated intravascular coagulation, renal failure, anuria or death in case of conflict in the ABO system,
allergic complications including anaphylactic shock | 15 days
  allergic complications including anaphylactic shock involving care in intensive care with intravenous injection of adrenaline, vis-à-vis precautions subsequent transfusions and biological investigations and immediate allergy and distance
infectious complications | 15 days
  infectious complications, including bacterial infections, viral, parasitic, including by poorly known or emerging agents
metabolic complications including febrile non-haemolytic reactions | 15 days
  metabolic complications including febrile non-haemolytic reactions, haemosiderosis and massive transfusion syndrome with hypocalcemia, acid-base imbalance, hyperkalemia, hemostasis disorders and hypothermia
lactate Rate | 15 days
central venous O2 saturation (SVO2) | 15 days
SOFA score (sepsis organ failure assessment) | 15 days
BNP Rate | 15 days
Death | 15 days
Cost reduction of transfusion | 15 days
  Cost reduction of transfusion support by reducing the number of PRBC transfusions, including costs related to medical and nursing time, biological examinations pre and post-transfusion, and packed red blood cells.
Rate of lactate | 15 days
  Rate of lactate
central venous O2 saturation (SVO2) | 15 days
  central venous O2 saturation (SVO2)
SOFA score (sepsis organ failure assessment) | 15 days
  SOFA score (sepsis organ failure assessment)
Rate BNP | 15 days
  Rate BNP

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abou Arab, Doctor, Principal Investigator — CHU Amiens-Picardie
Locations (2):
- France (2):
  - CHU Amiens Picardie, Amiens
  - Caen, Caen

REFERENCES:
- [Result] Fischer MO, Guinot PG, Debroczi S, Huette P, Beyls C, Babatasi G, Bafi K, Guilbart M, Caus T, Lorne E, Dupont H, Hanouz JL, Diouf M, Abou-Arab O. Individualised or liberal red blood cell transfusion after cardiac surgery: a randomised controlled trial. Br J Anaesth. 2022 Jan;128(1):37-44. doi: 10.1016/j.bja.2021.09.037. Epub 2021 Nov 30. PMID 34862002